CLINICAL TRIAL: NCT04698135
Title: Costituzione Della Biobanca Del Microbiota Intestinale e Salivare Umano: Dalla Disbiosi Alla Simbiosi
Brief Title: Establishment of the Human Intestinal and Salivary Microbiota Biobank - Obesity
Acronym: BIOMIS-Endo
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: University of Bari Aldo Moro (Other); University of Salento (Other); Istituti Tumori Giovanni Paolo II (Network); Institute of Biomembranes, Bioenergetics and Molecular Biotechnologies (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMIS-Endo
Record Dates: First submitted 2020-12-17; First posted 2021-01-06 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-01

CONDITIONS: Morbid Obesity; Metabolically Healthy Obesity
Keywords: Microbioma biobank; Biological human samples; obesity; Meta-omics approaches; Microbiota-pathology relationship
MeSH Terms: conditions — Obesity, Morbid; Obesity, Metabolically Benign; Obesity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — faeces, saliva, blood, serum, urine, PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- morbid obesity: Patients with morbid obesity
  Interventions: Other: Biological samples collection; Other: Questionnaire; Other: Medical/laboratory examinations
- Metabolically healthy obesity: Patients with metabolically healthy obesity
  Interventions: Other: Biological samples collection; Other: Questionnaire; Other: Medical/laboratory examinations
- Healthy volunteers: Healthy volunteers
  Interventions: Other: Biological samples collection; Other: Questionnaire; Other: Medical/laboratory examinations

INTERVENTIONS:
Other: Biological samples collection — Collection of faeces, coproculture examination, urine, saliva, PBMC and blood for biobanking, to evaluate the proteomic, metascriptomic, metabolomic, metagenomic, and metagenetic profile, and to perform routine screening. Analysis for the identification, quantification and characterization of health-promoting bacteria
Other: Questionnaire — Anamnestic questionnaire, 3-day food questionnaire, Food Frequency Questionnaire
Other: Medical/laboratory examinations — Blood pressure measurement, abdominal and thoracic physical examination, body composition through bioimpedance analysis and metabolic, cardiovascular and respiratory variables; OGTT 75gr for blood glucose and insulin at times 0, 30, 60, 90 and 120', and a nocturnal oximetry and subsequently, if necessary, overnight polysomnography for the diagnosis of obstructive sleep

SUMMARY:
This is a prospective, clinical, multicentre study aimed to collect biological samples and study microbiota from subjects with morbid obesity, metabolically healthy obesity and from healthy volunteers. Microbiota is a complex consortium of microorganisms, located at the mucosal level (in particular intestinal, oral and vaginal) having a key role in human health and in the onset of several diseases. Microbiota alterations have been found in several diseases (gastrointestinal, metabolic, renal, oncological, gynaecological)

The study will allow to:

* Provide biological samples (faeces, saliva, blood, urine) from healthy volunteers and patients to the first Italian microbiota biobank;
* Study microorganisms using different in vitro and in vivo techniques;
* Study the link between the microbiota and the disease. This study is part of the BIOMIS project (Project Code: ARS01_01220), presented as part of the "Avviso per la presentazione di progetti di ricerca industriale e sviluppo sperimentale nelle 12 aree di specializzazione individuate dal PNR 2015-2020" and admitted to funding under the National Operational Program "Ricerca e Innovazione" 2014-2020 by directorial decree of MIUR - Department for Higher Education and Research - n. 2298 of 12 September 2018. BIOMIS includes several clinical studies that enrol patients with different pathologies to collect and store biological samples and study microbiota.

DETAILED DESCRIPTION:
The primary aim of this multicentric study is to populate the first national microbioma biobank with biological samples (fecal, salivary, urinary and blood samples) subjects suffering from selected disease (morbid obesity, metabolically healthy obesity), and healthy volunteers.

The secondary aim is the characterization of microorganisms of the biobank and study of the microbiota-pathology relationship using meta-omics, in vitro and in vivo approaches.

The study plans to enrol 60 subjects at Policlinico of Bari, according to the inclusion/exclusion criteria. The study participation is voluntary, and the subjects have the right to withdraw from the study at any time and for any reason.

During the study, 3 visits are planned:

* Visit 0 (V0), including description of the objectives and procedures study, signature written informed consent, inclusion/exclusion criteria evaluation, medical examination (blood pressure measurement, abdominal and thoracic physical examination), body composition through bioimpedance analysis and metabolic, cardiovascular and respiratory variables; OGTT 75gr for blood glucose and insulin at times 0, 30, 60, 90 and 120', and a nocturnal oximetry and subsequently, if necessary, overnight polysomnography for the diagnosis of obstructive sleep, filling in of the anamnestic questionnaire, delivery of the coproculture kit, delivery of kits for the collection of fecal, salivary and urinary material to be reported at Visit 1 and delivery of a 3-day food diary, to be completed autonomously in the days preceding the Visit 1.
* Visit 1 (V1) - at least 4 days after V0, including delivery of the of the collected biological material (feces, saliva, urine), and of a 3-day food diary, filling in of the new signs and symptoms anamnestic questionnaire and blood sampling by medical staff.
* Telephone evaluation: administration of a "Food Frequency Questionnaire" to assess the subjects' alimentary habits.

Standard Operative Procedures (SOP) for samples storing, transport and processing will be adopted to ensure samples stability and grant results validity and quality.

Following collections, samples will be processed in different aliquots that will be used for:

* routine screening;
* storage in the first Italian human microbiote biobank (I.R.C.C.S. - Istituto Tumori "Giovanni Paolo II", Bari);
* evaluation of the proteomic, metascriptomic, metabolomic, metagenomic, and metagenetic profile;
* Evaluation of the transcriptomic profile of PBMCs of healthy subjects and subjects affected by selected pathologies and evaluation of the serum proteomic profile Furthermore, molecular characterization of pathogenic microorganisms and pathogenic biotypes (pathovars) of commensal species of subjects with selected pathologies will be conducted.

Part of the biological material will be used for animal studies on the physiopathological role of the human intestinal microbiota transplanted into mouse models of pathology and Germ-free mouse models (specific animal study protocol developed).

Also, in vitro studies on mucosal models to evaluate the interaction between the microbiota and the intestinal mucosa will be conducted.

The study foresees no more than minimal risk associated with blood sampling procedures. All the necessary measures to avoid any risks / inconveniences resulting from participation of the subject under study will be taken.

The study is compliant with Good Clinical Practice. Study protocol and all related documents have been approved by approved by the Independent Ethics Committees (IEC) of the involved clinical sites.

To ensure the protection and confidentiality of the participants' data, all study activities will be carried out in accordance with the European General Data Protection Regulation, Regulation (EU) 2016/679, which repeals Directive 95/46/EC.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY VOLUNTEERS

* healthy subjects aged between 18 and 60 years
* BMI between 18.5-30
* omnivorous diet
* signature of the informed consent

SUBJECTS WITH MORBID OBESITY

* subjects aged between 18 and 60 years
* subjects having morbid obesity (BMI ≥ 35 kg/m2), as following at least two of the following conditions: insulin resistance, prediabetes or type 2 diabetes mellitus, dyslipidemia, cardiovascular (arterial hypertension) and respiratory (obstructive sleep apnea) diseases
* omnivorous diet
* signature of the informed consent

SUBJECTS WITH METABOLICALLY HEALTHY OBESITY

* subjects aged between 18 and 60 years
* Obese subjects (BMI ≥ 35 kg/m2) metabolically healthy, without or with only one of the following : insulin resistance, prediabetes or type 2 diabetes mellitus, dyslipidemia, cardiovascular (arterial hypertension) and respiratory (obstructive sleep apnea) diseases
* omnivorous diet
* signature of the informed consent

  * Exclusion Criteria:

HEALTHY VOLUNTEERS/SUBJECTS WITH MORBID OBESITY/ METABOLICALLY HEALTHY OBESITY

* Current or previous infectious diseases (HAV, HBV, HCV, HIV, Cytomegalovirus, Epstein-Barr virus)
* Chronic liver disease
* History of Clostridium difficile infections
* Recent (<3 months) therapy with antibiotics, immunosuppressive drugs, chemotherapy
* Chronic therapy with proton pump inhibitors
* Recent (<3 months) use of probiotics, laxatives or other aids (drugs / supplements) for the regulation of gastrointestinal activity
* Previous history of organ / tissue transplantation
* Recent onset of diarrhea
* Chronic diarrhea
* Chronic constipation
* Previous gastrointestinal surgery (eg gastric bypass)
* Recurring urinary tract infections (3 cases per year)
* Previous major acute cardiovascular diseases (myocardial infarction, stroke)
* Type 2 diabetes mellitus
* Hypertension
* eGFR (estimated glomerular filtration rate) lower than 60ml / minute and / or diagnosis of nephropathy
* Chronic gastrointestinal disorders
* Systemic inflammatory diseases
* Suspicion, clinical diagnosis or previous history of cancer (<5 years)
* Autoimmune disorders or history of chronic and systemic autoimmune disorders
* Neurodegenerative disorders
* Pregnancy and breastfeeding
* Healthcare workers
* Operators work with animals
* Psychiatric conditions that reduce protocol compliance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with morbid obesity and metabolically healthy obesityattending one of the clinical centres involved in the study.
  Healthy volunteers will be recruited by invitation. Enrolled subjects must not have any family relationship and hierarchical subordination with the hospitals in which biological samples will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Biological samples collection for establishment of the first National Microbiome Biobank | through study completion, an average of 1 year
  Recruitment of 60 subjects (morbid obesity, metabolically healthy obesity and healthy volunteers) to collect biological samples for establishment of the first National Microbiome Biobank

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Giorgino, MD, Principal Investigator — Azienda Ospedaliera Universitaria Consorziale Policlinico di Bari
Locations (1):
- Azienda Ospedaliera Universitaria Policlinico di Bari - U.O.C. Endocrinologia Universitaria (D.E.T.O.), Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Z, Mocanu V, Cai C, Dang J, Slater L, Deehan EC, Walter J, Madsen KL. Impact of Fecal Microbiota Transplantation on Obesity and Metabolic Syndrome-A Systematic Review. Nutrients. 2019 Sep 25;11(10):2291. doi: 10.3390/nu11102291. PMID 31557953
- [Background] Aron-Wisnewsky J, Clement K, Nieuwdorp M. Fecal Microbiota Transplantation: a Future Therapeutic Option for Obesity/Diabetes? Curr Diab Rep. 2019 Jun 27;19(8):51. doi: 10.1007/s11892-019-1180-z. PMID 31250122
- [Background] Chen X, Devaraj S. Gut Microbiome in Obesity, Metabolic Syndrome, and Diabetes. Curr Diab Rep. 2018 Oct 18;18(12):129. doi: 10.1007/s11892-018-1104-3. PMID 30338410
- [Background] Kang Y, Cai Y. Gut microbiota and obesity: implications for fecal microbiota transplantation therapy. Hormones (Athens). 2017 Jul;16(3):223-234. doi: 10.14310/horm.2002.1742. PMID 29278509
- [Background] Marotz CA, Zarrinpar A. Treating Obesity and Metabolic Syndrome with Fecal Microbiota Transplantation. Yale J Biol Med. 2016 Sep 30;89(3):383-388. eCollection 2016 Sep. PMID 27698622